CLINICAL TRIAL: NCT03622970
Title: Video-Based Games for Upper Limb Rehabilitation in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Assist.Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108400987
Record Dates: First submitted 2018-07-22; First posted 2018-08-09 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VGBT with Nintendo® Wii and LMC games (Experimental): VGBT with Nintendo® Wii and LMC games:
  In order to improve the elbow and shoulder functions, Tennis and boxing, the games of Nintendo Wii® Fit WiiSports package that includes shoulder and elbow movements will be used for VGBT with Nintendo® Wii and Leap Motion Controller (LMC) games. In both of the games, the activities are carried out by providing feedback in the context of remote control and sound and vibration notifications.
  Interventions: Device: VGBT with Nintendo® Wii and LMC games
- NDT-based upper limb rehabilitation (Active Comparator): NDT-based upper limb rehabilitation:
  NDT-based upper limb rehabilitation aims to facilitate normal movement for upper extremity activities such as getting dressed and eating etc by using real materials (clothes, spoons, pencils, buttons, rope, etc.). The target activities were practised with the materials such as velcro cylinders, skill cubes, exercise bands, screw sets, therapeutic putty, and tripled coordination tools.
  Interventions: Behavioral: NDT-based upper limb rehabilitation

INTERVENTIONS:
Device: VGBT with Nintendo® Wii and LMC games — Nintendo Wii and LMC games will be used for upper limb rehabilitation in Cerebral Palsy. The games are tennis and boxing for Nintendo Wii, Leapball and CatchApet for LMC.
  Arms: VGBT with Nintendo® Wii and LMC games
Behavioral: NDT-based upper limb rehabilitation — NDT-based upper limb rehabilitation includes using real materials (clothes, spoons, pencils, buttons, rope, etc.) such as getting dressed and eating etc. Also, It will practised with the materials such as velcro cylinders, skill cubes, exercise bands, screw sets, therapeutic putty, and tripled coordination tools.
  Arms: NDT-based upper limb rehabilitation

SUMMARY:
The aim of the present study is to compare the effects of Neurodevelopmental Treatment (NDT)-based upper limb rehabilitation and video-game based therapy (VGBT) with Nintendo® Wii and LMC games on upper extremity functions in patients with Cerebral Palsy (CP).

DETAILED DESCRIPTION:
The investigators hypothesized that VGBT using the Nintendo® Wii and LMC would be a usable tool to train manual dexterity in patients with CP as comprehensive and holistic therapy.

The NDT program for both groups will be routinely applied according to each child's individual needs and included tonus regulation, support of sensation, perception and motor development for gross motor function.

The two different patient-centered rehabilitation programs will be conducted with an average of one hour sessions three times a week for 8 weeks in both groups. The two different patient-centered programs will be as VGBT with Nintendo® Wii and LMC games (Group I) and NDT-based upper limb rehabilitation (Group II).

ELIGIBILITY:
Inclusion Criteria:

The health committee report has received a CP diagnosis

* Being between 5-18 years of age
* According to Modifiye Ashworth Scale (MAS), upper extremity spasticity (0), (1), (1+)
* Ability to adapt to exercises (According to the health report mental level normal or "mild mental retardation"

Exclusion Criteria:

* Botulinium Toxin (BOTOX) injection for the upper extremity in the last 6 months
* Does not have epileptic epilepsy
* Any person who has been diagnosed as having any absence of a cardiac or orthopedic condition
* Admission of family treatment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Minnesota Hand Dexterity Test | Change from baseline to 8 weeks, follow up at two months
  Minnesota Manual Dexterity Test (MMDT): is a short version of the Minnesota Dexterity Tests and consists of two timed sub-tests ("placing" and "turning tests") to assess the required manual dexterity to turn and/or place 60 short, round blocks with one or both hands . In this study, the placing sub-test will be used to assess the ability to handle objects, measured by the time required to complete the task.

SECONDARY OUTCOMES:
Modified Ashworth Scale | Change from baseline to 8 weeks, follow up at two months
  Modified Ashworth Scale (MAS) measures the muscle spasticity rate (score, 0-5). Spasticity of wrist flexors, elbow flexors and forearm pronators will be assessed due to MAS in this study. Participants sat with their forearm fully supported and will be instructed to relax. The measurer moves the wrist into extension as fast as possible and then rated the quality of the muscle reaction to stretch on a scale from 0 to 5, with 0 representing no spasticity.
Hand and pinch grips | Change from baseline to 8 weeks, follow up at two months
  Grip strength was measured using a standard adjustable handle Jamar® Plus+Hand Dynamometer (Irvington NY, USA) in the sitting position with the shoulder adducted and neutrally rotated and the elbow flexed at 90. Pinch strengths (tip, key and palmar pinch) will be measured by a hydraulic pinch gauge (Irvington NY, USA) in the sitting position with the shoulder adducted and neutrally rotated and the elbow flexed at 90. Pinch positions will be defined using the American Society for Hand Therapists guideline. Each of grip and pinch strength tests will be performed thrice with a 30-sec interval between tests, and the mean value will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided